CLINICAL TRIAL: NCT00476645
Title: Fulvestrant in Hormone-refractory Prostate Cancer
Brief Title: Fulvestrant in Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-01890; 96025 (Other: Stanford University alternate IRB Number); PROS0010 (Other: OnCore)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fulvestrant (Experimental)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 250 mg IM on Days 1 and 14 in the first month, thereafter 250 mg monthly
  Other Names: Faslodex; ICI 182,780

SUMMARY:
The purpose of this study is to determine if treatment with fulvestrant leads to a slowing of tumor progression in patients who have developed androgen-independent (AIPC) or hormone-refractory prostate cancer (HRPC) and who have a rising serum prostate specific antigen (PSA).

DETAILED DESCRIPTION:
The purpose of this study is to determine if treatment with fulvestrant leads to a slowing of tumor progression in patients who have developed androgen-independent (AIPC) or hormone-refractory prostate cancer (HRPC) and who have a rising serum prostate specific antigen (PSA). In vitro studies have shown that fulvestrant downregulates androgen receptor (AR) in LNCaP cancer cell lines to a significant extent, thereby inhibiting growth of tumor cells. In addition, it is important to emphasize that fulvestrant has also been found to decrease growth of AR-negative prostate cancer cells. These observations provide the rational for using fulvestrant for the treatment of AIPC and HRPC.

ELIGIBILITY:
Inclusion Criteria:

* Must give signed written informed consent
* Must be of age 18 years or older
* Histologically confirmed adenocarcinoma of the prostate
* Must be currently receiving LHRH agonists and have castrate levels of testosterone or have had an orchiectomy
* Must have had rise in PSA despite anti-androgen withdrawal
* Must exhibit two consecutive rises in PSA after the last hormonal manipulation
* Minimum PSA > 5mg/dL
* KPS > 80%
* Up to one prior chemotherapy treatments allowed
* Life expectancy of greater than 6 months

Exclusion Criteria:

* Concomitant hormonal therapy other than an LHRH
* Noncompliance
* Platelets less than 100 x 10e9 /L
* International normalization ratio (INR) greater than 1.6
* Total bilirubin greater than 1.5 x ULRR
* ALT or AST greater than 2.5 x ULRR if no demonstrable liver metastases or greater than 5.0 x ULRR in presence of liver metastases
* History of bleeding diathesis (ie, disseminated intravascular coagulation [DIC], clotting factor deficiency)
* History of long-term anticoagulant therapy (other than antiplatelet therapy)
* History of hypersensitivity to active or inactive excipients of fulvestrant (ie, castor oil or Mannitol)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Srinivas S, Harshman LC, Feldman D. "Effect of fulvestrant on PSA doubling time in patients with castration-resistant prostate cancer (CRPC)." JCO. Annual Meeting, ASCO 2010. 20 May 2010;28(15-suppl)(abs e15112).

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant 250 mg: IM fulvestrant (250 mg) day 1 & day 14 of 1st month, then monthly
Period: Overall Study
Arm/Group | Fulvestrant 250 mg
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis
Arm/Group | Fulvestrant 250 mg
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 75 [58 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: PSA Reduction ≥ 50%
Description: Number of subjects with serum PSA reduction ≥ 50% at 3 months
Time Frame: 3 months
Population: All subjects (10 males) had castration-resistant prostate cancer. 6 had recieved prior radical prostatectomy as primary therapy. 4 had received prior chemotherapy. The majority had previously received 2 hormonal therapies. 2 had recieved radiation therapy, and 2 had recieved hormonal monotherapy.
Measure: Number; unit: participants
Arm/Group | Fulvestrant 250 mg
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: PSA Doubling Time
Description: Number of subjects with prolongation of PSA doubling time
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Fulvestrant 250 mg
Number analyzed (Participants) | 10
participants | 3

3. Secondary Outcome: Stable Disease After One Year
Description: Stable disease was defined as continuing treatment without disease progression, with disease progression defined as 3 consecutive rises in serum PSA or objective progression by RECIST criteria.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Fulvestrant 250 mg
Number analyzed (Participants) | 10
participants | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Fulvestrant 250 mg
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 250 mg (N=10)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Edema (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Intermittent tiny sensitive area on forehead (sligh (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No